CLINICAL TRIAL: NCT00512226
Title: Clinical and Laboratory Assessment of Iron Overload in Sickle Cell Anemia and Sickle Cell Thalassemia Using T2* Cardiac MRI.
Brief Title: Iron Overload Assesment in Sickle Cell Anemia and Sickle Cell Thalassemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0037-07-EMC
Record Dates: First submitted 2007-08-05; First posted 2007-08-07 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Sickle Cell Anemia; Sickle Cell Thalassemia; Iron Overload; MRI
Keywords: Sickle Cell Anemia; Sickle Cell Thalassemia; Iron Overload; MRI
MeSH Terms: conditions — Anemia, Sickle Cell; Iron Overload

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cardiac and Liver T2* MRI — Laboratory examinations that are routinely used in follow up of those patients and T2* MRI analysis.

SUMMARY:
Iron overload is well study in Thalassemia patients and it's not only related to blood transfusions, since intestinal iron absorption is also increased in those patients. Sickle cell patients didn't develope significant clinical symptoms and signs of iron overload in spite frequent transfusions. The purpouse of this study is to assess the iron overload in Sickle cell anemia and Sickle cell Thalassemia patients using clinical parameters and cardiac T2*MRI in order to determine the cardiac and liver iron.

ELIGIBILITY:
Inclusion Criteria:

* All the patients with Sickle cell anemia and Sickle cell Thalasemia that are currently in follow up at the Pediatric Hematology Unit

Exclusion Criteria:

* Age below 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Assessment of Iron overload. | December 2008

SECONDARY OUTCOMES:
Institute the criteria for iron chelator treatment | December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Principal Investigator — Pediatric Hematology Unit, Ha'Emek Medical Center
Locations (1):
- Pediatric Hematology Unit and Pediatric Dpt B - HaEmek Medical Center, Afula, Israel